CLINICAL TRIAL: NCT05555030
Title: iCura Diagnostics, LLC / COVID-19 Antigen Rapid Home Test Over the Counter Rapid Antigen Self-Test for Detection of SARS-CoV-2 Virus: Clinical Evaluation
Brief Title: COVID-19 iCura SARS-CoV-2 Ag OTC: Clinical Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Day Diagnostics (Network)
Collaborators: Paragon Rx Clinical, Inc. (Unknown); iCura Diagnostics, LLC (Unknown)
Responsible Party: Principal Investigator, Jason Liggett, Chief Scientist, New Day Diagnostics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDP-OTC-iCD-001
Record Dates: First submitted 2022-09-12; First posted 2022-09-26 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: SARS-CoV-2 Infection; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is an open-label, prospective study to evaluate the sensitivity and specificity of the iCura COVID-19 Antigen Rapid Home Test when a lay person conducts the test on themselves or another study participant. Potential subjects will be those presenting for COVID-19 testing. The study will evaluate the performance of the iCura COVID-19 Antigen Rapid Home Test by comparing it to a high sensitivity EUA SARS-CoV-2 RT-PCR assay to calculate both the positive percent agreement (PPA, or sensitivity) and the negative percent agreement (NPA, or specificity).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- At least 30 children between 2 and 13 years of age (Experimental): Participants 2-13 years of age will have a nasopharyngeal swab sample collected by trained study site personnel for testing on a high sensitivity EUA SARS-CoV-2 RT-PCR assay to compare the result to the result of the iCura SARS-CoV-2 Antigen Rapid Home Test. The parent or legal guardian of the child will collect an anterior nasal swab sample from the child and perform the iCura SARS-CoV-2 Antigen Rapid Home Test.
  Interventions: Device: iCura COVID-19 Antigen Rapid Home Test; Diagnostic Test: RT-PCR Test
- Subject 14-65+ years of age (Experimental): Participants will have a nasopharyngeal swab sample collected by trained study site personnel for testing on a high sensitivity EUA SARS-CoV-2 RT-PCR assay to compare the result to the result of the iCura SARS-CoV-2 Antigen Rapid Home Test. The participant will then self-collect or, if both are over 18, collect from another study participant an anterior nasal swab sample and test using the iCura SARS-CoV-2 Antigen Rapid Home Test.
  Interventions: Device: iCura COVID-19 Antigen Rapid Home Test; Diagnostic Test: RT-PCR Test

INTERVENTIONS:
Device: iCura COVID-19 Antigen Rapid Home Test — Candidate Ag self-test kit anterior nasal specimen collection and testing will be done under the supervision of qualified site personnel in person. Comparator NP samples shall be collected at least 15 minutes prior to Ag samples with at least 15 minutes between nasal collections including collections that may occur prior to study enrollment. Comparator samples will be collected first by qualified personnel at a study site or physician's office using an FDA authorized nasopharyngeal swab collection kit and SARS-CoV-2 molecular assay.
Diagnostic Test: RT-PCR Test — High sensitivity RT-PCR COVID-19 Test

SUMMARY:
SARS-CoV-2 rapid antigen over the counter clinical performance evaluation.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) is a disease caused by a newly discovered coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)1. The SARS-CoV-2 is a β-coronavirus, which is enveloped non-segmented positive-sense RNA virus 22. It is spread by human-to-human transmission via droplets or direct contact, and infection has been estimated to have mean incubation period of 6.4 days and a basic reproduction number of 2.24-3.58. Among patients with pneumonia caused by SARS-CoV-2, fever was the most common symptom, followed by cough. On 11 March 2020, the COVID-19 outbreak was characterized as a pandemic by the WHO. Since then, over 70 million people worldwide have been infected with the virus with over 1.5 million deaths attributed to the virus5. Laboratory testing for SARS-CoV-2 is currently being performed to determine if an individual has active infection via detection of viral RNA or if an individual has an immune response to the virus from a previous infection via detection of antibodies.

Specimen collection is a crucial first step in the evaluation of an individual's SARS-CoV-2 infection status. The goal of this project is to evaluate a Candidate Ag self-test kit for over the counter (OTC) use. Study subjects under EDP supervision, either in-person or via video conference, will collect and test anterior nasal swab samples and a Study Representative will collect and ship a nasopharyngeal swab sample for comparator PCR testing. The Candidate Ag self-test kit collection and testing methodology is viewed as a convenient and inexpensive method to test clinical specimens for SARS-CoV-2 and OTC access will improve the availability of COVD-19 testing.

The iCura COVID-19 Antigen Rapid Home Test (candidate test) is a rapid antigen (Ag) immunochromatography based one step in vitro test intended to detect nucleocapsid antigen from the SARS-CoV-2 virus that causes COVID-19. It is designed for over the counter (OTC) rapid qualitative determination of SARS-CoV-2 virus antigen in anterior nasal swabs from individuals within 14 days of symptom onset or without symptoms or other epidemiological reasons to suspect COVID-19 infection. This test is for non-prescription home use with self-collected anterior nasal swab specimens directly from individuals aged 14 years and older or with adult-collected anterior nasal samples directly from individuals aged 2 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Lay subjects greater than 2 years old that do not know their current COVID-19 status and can complete the consent/assent process in both written and spoken English may be included in the study.

Exclusion Criteria:

* Subjects less than 2 years old will be excluded.
* Participants that are or were medial and/or laboratory professionals will be excluded.
* Participants that cannot read and understand English will be excluded.
* High risk individuals will not be excluded unless they are too young or have prior training or experience that would exclude them.
* Participants who refuse to sign the informed consent/assent form(s) will be excluded.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Positive Percent Agreement | 3 months
  The acceptance criteria for this study is Positive Percent Agreement (PPA) greater than or equal to eighty percent in a comparison between the iCura COVID-19 Antigen Rapid Home TestRT-PCR comparator test results
Negative Percent Agreement | 3 months
  The acceptance criteria for this study is a Negative Percent Agreement (NPA) greater than or equal to ninety-eight percent in a comparison between the iCura COVID-19 Antigen Rapid Home Test and the RT-PCR comparator test results.

SECONDARY OUTCOMES:
Detection of Asymptomatic Positives | 3 months
  Number of participants with a positive PCR comparator result, but reported no symptoms or epidemiological reasons to suspect COVID-19 infection within the past 14 days. This will be compared to their iCura COVID-19 Antigen Rapid Home Test result to determine the ability of the iCura COVID-19 Antigen Rapid Home Test to detect individuals who are infected but are not symptomatic.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Liggett, PhD, Principal Investigator — New Day Diagnostics
Locations (2):
- United States (2):
  - Paragon, Anaheim, California
  - EDP Biotech, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119
- [Background] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- See also: WHO. 2022 — https://www.who.int/
- See also: Johns Hopkins University Center for Health Security Website. 2020 — https://www.centerforhealthsecurity.org